CLINICAL TRIAL: NCT05047731
Title: Antihypertensive Deprescribing in Long-term Care: A Randomized Controlled Trial (OptimizeBP)
Brief Title: Antihypertensive Deprescribing in Long-term Care
Acronym: OptimizeBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00097312
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Frailty
Keywords: Pragmatic trial; Long-term care; Nursing home; Hypertension; Antihypertensive agents; Deprescriptions; Routinely collected health data; Frail older adult
MeSH Terms: conditions — Hypertension; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deprescribing group (Experimental): The facility pharmacist will actively deprescribe antihypertensive medication of residents in this group.
  Interventions: Drug: Antihypertensive medication
- Usual care group (No Intervention): The facility pharmacist and the attending physician will provide usual care to residents in this group, and this includes quarterly medication reviews.

INTERVENTIONS:
Drug: Antihypertensive medication — Antihypertensive medication will be continually reduced provided an upper systolic threshold of 145 mmHg is not exceeded
  Arms: Deprescribing group

SUMMARY:
Frail older adults are commonly prescribed blood pressure medication, yet it is unclear if blood pressure medication is actually beneficial for them. Observational studies in this population suggest blood pressure medication has limited benefit and may even be harmful, including an increased risk for falls and cognitive impairment. Randomized controlled trials are needed to confirm this.

This study is a randomized controlled trial of blood pressure medication deprescribing, amongst long-term care residents with systolic blood pressure lower than 135 mmHg. In the intervention group, with physician consent, the facility pharmacist or nurse practitioner will continually reduce antihypertensives provided an upper systolic threshold of 145 mmHg is not exceeded. The control group will receive usual care. The hypothesis is that avoiding unnecessarily low systolic blood pressure is beneficial in a frail, end-of-life population.

DETAILED DESCRIPTION:
Observational evidence suggests antihypertensive medications have limited benefit and may even be harmful in the frail older adult population. Although more modest blood pressure targets are already recommended, the impact of deprescribing antihypertensive medication on mortality and morbidity in the frail older adult population has yet to be confirmed by randomized controlled trials.

The objective of this study is to determine, in hypertensive long-term care residents with a systolic blood pressure below 135 mmHg, whether "deprescribing" antihypertensive medications (provided an upper systolic threshold of 145 mmHg is not exceeded), compared to no change in prescribing, will delay all-cause mortality (our primary outcome).

The study is an event-driven 2-parallel group randomized controlled trial, to be conducted in participating Alberta long-term care (LTC) facilities. The trial operates under a waiver of consent, as the intervention is recommended care, with residents, physicians, and family having the ability to opt individual residents out of the study before eligibility is determined. Eligibility will be determined using linked administrative claims databases holding physician diagnoses and medication dispensed, and by using usual care systolic blood pressure collected by the LTC facility. The provincial data steward (Alberta Health Services) will access this data, determine eligibility, individually randomize eligible residents who have not opted out, and advise the facility pharmacist which patients are in the intervention group.

Facility pharmacists or nurse practitioners will then stop or reduce doses of antihypertensive medication in the intervention group according to a pre-defined deprescribing algorithm. The data steward will track outcomes using administrative claims data, and the study will end once 247 primary outcome events have been observed. This is anticipated to occur 3-years post the start of randomization. An interim data safety monitoring board, chaired by Dr. James M.Wright, hypertension specialist and Co-ordinating Editor of the Cochrane Hypertension Review Group, will convene upon observing 124 primary outcomes. This group will recommend whether or not the study should stop early based on observed efficacy, or safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* ≥2 diagnoses (dx) of hypertension from either a community practitioner or/and from a hospital admission.
* On ≥1 oral antihypertensive medication (requires a dispensation in the preceeding 15 days).
* Average recorded systolic BP of <135 mmHg.

Exclusion Criteria:

* ≥2 community dx of congestive heart failure, ≥1 dx of in hospital congestive heart failure, ≥1 dx of emergency visit of congestive heart failure, dx of congestive heart failure in RAI-MDS 2.0, or prescription of furosemide in the last 15 days.
* The resident's only antihypertensive prescribed is a beta blocker.
* The resident's only antihypertensive prescribed is a calcium channel blocker and the resident has ≥1 health system encounters with a diagnosis of angina.
* The resident's only antihypertensive prescribed is an alpha blocker.
* Admitted to the hospital at the time of randomization; or opted out of the trial by the resident, their family, their physician, or the facility.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 522 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  All-cause death - as recorded in government health claim databases

SECONDARY OUTCOMES:
Composite of All-Cause Mortality or All-Cause Unplanned Hospitalization | through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  Composite of all-cause death and unplanned hospital admission or emergency room visit - as recorded in government health claim databases

OTHER OUTCOMES:
All-Cause Unplanned Hospitalization | through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  All cause hospitalization or emergency room visit excluding elective surgeries or booked procedures/planned follow-up care - as recorded in governmental health claims databases
Non-Vertebral Fracture | through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  Any physician billing (hospital or community) for a fracture other than a vertebral fracture (which might indicate a vertebral compression fracture secondary to osteoporosis, and not trauma) - as recorded in government health claim databases
Number of Participants with Record of ≥1 Fall in Last 30-days | 4.5 Months (average - will occur within a 3- to 6-month post randomization window)
  As recorded in the first quarterly Resident Assessment Instruction Minimum Data Set 2.0 (RAI-MDS 2.0) at the LTC facility in the 3- to 6-month window following randomization
Number of Participants with Partial or Full Thickness Skin Ulceration (stage 2 to 4) | 4.5 Months (average - will occur within a 3- to 6-month post randomization window)
  As recorded in the first quarterly RAI-MDS 2.0 assessment at the LTC facility in the 3- to 6-month window following randomization
Number of Participants with Renal Insufficiency | ≥6-weeks post-randomisation through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  Any eGFR <30 ml/min/1.73m2 ≥6-weeks post-randomisation as recorded in governmental health claim databases
Unplanned All-Cause Hospitalization with a Diagnosis of Stroke, Heart Attack, Congestive Heart Failure or Atrial Fibrillation | through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  Unplanned hospital admission or emergency room visit for stroke, acute coronary syndrome/myocardial infarction, heart failure, or atrial fibrillation - as recorded in governmental health claims databases
Number of Participants with "Deteriorated Cognition as Compared to Status 90 Days Prior" | 4.5 Months (average - will occur within a 3- to 6-month post randomization window)
  As recorded in the first quarterly RAI-MDS 2.0 at the LTC facility in the 3- to 6-month window following randomization
Number of Participants with "Deteriorated Mood as Compared to Status 90 Days Prior" | 4.5 Months (average - will occur within a 3- to 6-month post randomization window)
  As recorded in the first quarterly RAI-MDS 2.0 assessment at the LTC facility in the 3- to 6-month window following randomization
Number of Participants with "Deteriorated Activities of Daily Living (ADL) as Compared to Status 90 Days Prior" | 4.5 Months (average - will occur within a 3- to 6-month post randomization window)
  As recorded in the first quarterly RAI-MDS 2.0 assessment at the LTC facility in the 3- to 6-month window following randomization
Number of Participants with "Behavioural Symptoms that are Present a Minimum of 4 Days per Week and Not Easily Altered" Including a) Wandering, b) Verbal Abuse, c) Physical Abuse, d) Socially Inappropriate or Disruptive Behaviour, or e) Resisting Care | 4.5 Months (average - will occur within a 3- to 6-month post randomization window)
  As recorded in the first quarterly RAI-MDS 2.0 assessment at the LTC facility in the 3- to 6-month window following randomization
Acute Care Costs | through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  Calculated from each hospital/emergency admission's resource intensity weight as recorded in government health claim databases
Total Costs of Care | through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  Acute care costs + medication costs + physician billings + nursing/facility costs as recorded in governmental health claims data. Nursing/facility costs will be estimated from level of care and duration of stay.
Number of Antihypertensive Medications with ≥25%, ≥50%, and 100% Reduction from Baseline in Dosage Dispensed | 3- and 6-months post-randomization
  As recorded in government health claim databases
Number of Participants with ≥1 Baseline Antihypertensive Medication with ≥25%, ≥50%, and 100% Reduction in Dosage Dispensed | 3- and 6-months post-randomization
  As recorded in government health claim databases
Number of Participants with the Addition of ≥1 New Antihypertensive Medication or Increase in Dosage from Baseline. | 3- and 6-months post-randomization
  As recorded in government health claim databases
Number of Discrete Antihypertensive Medications Used in the Last 15 days (baseline, 3- and 6-months post-randomisation) | 3- and 6-months post-randomization
  As recorded in government health claim databases
Number of Discrete Medications Used in the Last 15 Days (baseline, 3- and 6-months post-randomisation) | 3- to 6-months post-randomization
  As recorded in government health claim databases
Average Systolic Blood Pressure and Average Diastolic Blood Pressure | through study completion (estimated to be 4 years, trial will continue until 247 participants have experienced the primary outcome event)
  As recorded by the long-term care facility

CONTACTS AND LOCATIONS:
Overall Officials: Roni Kraut, Principal Investigator — University of Alberta
Locations (1):
- Multiple long-term care facilities, Multiple Locations, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Although we hope to make a de-identified participant-level version of our final analytic dataset publicly available on our website (www.PragmaticTrials.ca), and will request to do so, this requires the permission of Alberta Health Services, who must weigh the privacy concerns.
Supporting Information: Study Protocol, SAP
Time Frame: If approval from Alberta Health Services is obtained, data will be posted co-incident with the main results publication and intended for long-term availability.
Access Criteria: The data will be downloadable in the form of an Excel spreadsheet for anyone who wishes to access it. No application process will be necessary.
URL: https://pragmatictrials.ca/

REFERENCES:
- [Result] Kraut RY, Youngson E, Sadowski CA, Bakal JA, Faulder D, Korownyk CS, Vucenovic A, Eurich DT, Manca DP, Lundby C, Kivi P, Manville M, Garrison SR. Antihypertensive deprescribing in frail long-term care residents (OptimizeBP): protocol for a prospective, randomised, open-label pragmatic trial. BMJ Open. 2024 Aug 29;14(8):e084619. doi: 10.1136/bmjopen-2024-084619. PMID 39209778
- See also: OptimizeBP protocol — https://bmjopen.bmj.com/content/14/8/e084619